CLINICAL TRIAL: NCT01594281
Title: Multicenter Randomized Open-label Three-arms Controlled 12 Months Clinical Proof of Concept Study to Evaluate Efficacy and Safety of Ranibizumab Alone or in Combination With Laser Photocoagulation vs. Laser Photocoagulation Alone in Proliferative Diabetic Retinopathy
Brief Title: Multicenter 12 Months Clinical Study to Evaluate Efficacy and Safety of Ranibizumab Alone or in Combination With Laser Photocoagulation vs. Laser Photocoagulation Alone in Proliferative Diabetic Retinopathy (PRIDE)
Acronym: PRIDE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRFB002DDE21; 2011-005542-35 (EudraCT Number)
Record Dates: First submitted 2012-05-03; First posted 2012-05-09 (Estimated); Results first posted 2019-03-15 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2018-11

CONDITIONS: Proliferative Diabetic Retinopathy (PDR)
Keywords: Panretinal photocoagulation; Ranibizumab
MeSH Terms: interventions — Ranibizumab

STUDY DESIGN:
Masking Description: An open-label design was chosen in which the evaluation of the primary objective was performed by a reading center. The reading center that evaluated the primary and several secondary objectives was blinded to randomization and therefore assessed these objectives uninfluenced by treatment information. However, laser burns were visible on the images, and no full blinding regarding panretinal laser photocoagulation (PRP) was possible for the reading center.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ranibizumab mono (Experimental): Interventional Core Phase: One intravitreal injection of ranibizumab 0.5 mg to the study eye monthly until stability regarding morphological parameters is confirmed (ie, no further improvement of morphology or no worsening of morphology for 3 consecutive months)
  Interventions: Drug: Ranibizumab 0.5 mg
- PRP mono (Active Comparator): Interventional Core Phase: Panretinal laser photocoagulation (PRP) treatment administered to the study eye in accordance with the modified diabetic retinopathy study (DRS) guidelines for panretinal laser photocoagulation procedures
  Interventions: Procedure: Panretinal laser photocoagulation
- Ranibizumab+PRP (Experimental): Interventional Core Phase: Ranibizumab 0.5 mg as described for the ranibizumab mono arm and PRP treatment as described for the PRP mono arm until stability regarding morphological parameters is confirmed
  Interventions: Drug: Ranibizumab 0.5 mg; Procedure: Panretinal laser photocoagulation

INTERVENTIONS:
Drug: Ranibizumab 0.5 mg — Pre-filled syringe for intravitreal injection
  Other Names: Lucentis®; RFB002
  Arms: Ranibizumab mono; Ranibizumab+PRP
Procedure: Panretinal laser photocoagulation — PRP treatment following DRS guidelines
  Other Names: PRP
  Arms: PRP mono; Ranibizumab+PRP

SUMMARY:
The purpose of this study was to assess the efficacy and safety of the anti-Vascular Endothelial Growth Factor (VEGF) agent ranibizumab (0.5 mg) with or without Panretinal laser photocoagulation (PRP) compared to PRP alone in patients with Proliferative Diabetic Retinopathy (PDR).

DETAILED DESCRIPTION:
A 12-month core phase was followed by a 12-month observational follow-up phase (physician's routine), for a planned individual study duration of 24-25 months. A separate informed consent was signed for the 12-month observational follow-up phase. This study was conducted in Germany.

ELIGIBILITY:
Inclusion Criteria:

* Proliferative Diabetic Retinopathy
* Best Corrected Visual Acuity (BCVA) in study eye of at least 20 Early Treatment Diabetic Retinopathy Study (ETDRS) letters (20/400)
* Type 1 or type 2 diabetes under medical surveillance / with stabilized treatment

Exclusion Criteria:

* Proliferative vitreoretinopathy in study eye
* Clinically significant macular edema (CSME) in the study eye
* Clinically non significant macular edema (CNSME) that is likely to develop to CSME in the study eye
* Uncontrolled glaucoma in either eye
* Other protocol-specified conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2012-12-11 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2017-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (21):
- Germany (21):
  - Novartis Investigative Site, Aachen
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Darmstadt
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Glauchau
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hösbach
  - Novartis Investigative Site, Karlsruhe
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Marburg
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Regensburg
  - Novartis Investigative Site, Tübingen
  - Novartis Investigative Site, Ulm

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were screened for eligibility at 23 German study sites and randomized at 22 of the 23 sites.
Pre-assignment Details: The number of patients in the protocol section (107) excludes one patient in the Ranibizumab mono arm who withdrew prior to the baseline visit. The number of patients in the Randomized Set (108) includes this patient. A separate Informed Consent was signed for the Non-Interventional Follow Up Phase
Groups:
- Ranibizumab Mono: Interventional Core Phase: One intravitreal injection of ranibizumab 0.5 mg to the study eye monthly until stability regarding morphological parameters is confirmed (ie, no further improvement of morphology or no worsening of morphology for 3 consecutive months)
  Non-interventional Follow-Up Phase: Treatment per physician´s routine standard of care until Month 24
- PRP Mono: Interventional Core Phase: Panretinal laser photocoagulation (PRP) treatment administered to the study eye in accordance with the modified diabetic retinopathy study (DRS) guidelines for panretinal laser photocoagulation procedures. If stability of morphological parameters could not be confirmed after 3 months, additional laser treatment was initiated.
  Non-Interventional Follow-Up Phase: Treatment per physician´s routine standard of care until Month 24.
- Ranibizumab+PRP: Interventional Core Phase: Ranibizumab 0.5 mg as described for the ranibizumab mono arm and PRP treatment as described for the PRP mono arm until stability regarding morphological parameters is confirmed
  Non-interventional Follow-Up Phase: Treatment per physician´s routine standard of care until Month 24
Period: Interventional Core Phase
Arm/Group | Ranibizumab Mono | PRP Mono | Ranibizumab+PRP
Started (All randomized patients, including one patient who withdrew prior to the baseline visit) | 36 | 36 | 36
Full Analysis Set (FAS) (All randomized patients with at least one study treatment and one post-baseline assessment) | 35 | 35 | 36
Completed (End of Core Study (EOCS), defined as the last visit under therapy, up to Month 12) | 29 | 26 | 28
Not Completed | 7 | 10 | 8
Not completed — Protocol Deviation | 1 | 0 | 0
Not completed — Subject Withdrew Consent | 0 | 1 | 1
Not completed — Death | 1 | 1 | 2
Not completed — Lost to Follow-up | 1 | 4 | 1
Not completed — Adverse Event | 4 | 4 | 4
Period: Non-Interventional Follow Up Phase
Arm/Group | Ranibizumab Mono | PRP Mono | Ranibizumab+PRP
Started (All patients signing an Informed Consent, including one patient who withdrew without documented data) | 28 (1 patient exited after completing Core Phase and did not start the Follow-Up Phase) | 21 (5 patients exited after completing Core Phase and did not start the Follow-Up Phase) | 25 (3 patients exited after completing Core Phase and did not start the Follow-Up Phase)
Follow Up Set (FUS) (All patients with documented data in the follow up phase) | 28 | 20 | 25
Completed | 25 | 19 | 23
Not Completed | 3 | 2 | 2
Not completed — Lost to Follow-up | 2 | 2 | 0
Not completed — Administrative Problems | 0 | 0 | 1
Not completed — Subject Withdrew Consent | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Set
Groups:
- Total: Total of all reporting groups
Arm/Group | Ranibizumab Mono | PRP Mono | Ranibizumab+PRP | Total
Number analyzed (Participants) | 35 | 35 | 36 | 106
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.5 (11.0) | 53.0 (12.1) | 55.0 (13.4) | 53.5 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 11 | 8 | 33
  Male | 21 | 24 | 28 | 73
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Area of Neovascularizations (NVs) at End of Core Study (EOCS)
Description: The area of neovascularizations (NV) was assessed by a central reading center via fluorescein angiography (FA) images. The area of NV was calculated as the sum of area of neovascularization of the disc (NVD) and neovascularization elsewhere (NVE) and was recorded in square millimeters. A higher positive change value may indicate a greater formation of new, abnormal blood vessels and thus disease progression. One eye (study eye) contributed to the analysis.
Time Frame: Baseline, EOCS
Population: FAS; LOCF. Only patients with both values at baseline and any post-baseline value were included.
Measure: Mean (Standard Deviation); unit: square millimeters
Arm/Group | Ranibizumab Mono | PRP Mono | Ranibizumab+PRP
Number analyzed (Participants) | 33 | 33 | 33
square millimeters | -4.6 (11.3) | -0.9 (3.9) | -1.7 (3.0)
Statistical Analysis 1: Comparison: Ranibizumab Mono vs PRP Mono; Test type: Other — The focus of this PoC study was not on hypothesis testing but on a rough estimation of differences between treatments. The usual p-values are provided as a descriptive tool; p = 0.0344, ANCOVA; Least Squares Mean Difference = -2.8, 95% CI 2-sided [-5.4 to -0.2]
Statistical Analysis 2: Comparison: Ranibizumab Mono vs Ranibizumab+PRP; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.3809, ANCOVA; Least Squares Mean Difference = -1.2, 95% CI 2-sided [-3.8 to 1.5]
Statistical Analysis 3: Comparison: PRP Mono vs Ranibizumab+PRP; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.2113, ANCOVA; Least Squares Mean Difference = 1.7, 95% CI 2-sided [-1.0 to 4.3]

2. Secondary Outcome: Change From Baseline in Area of Neovascularizations (NVs) at Month 3
Description: as for outcome 1
Time Frame: Baseline, Month 3
Population: FAS; LOCF. Only patients with both values at baseline and any post-baseline value were included.
Measure: Mean (Standard Deviation); unit: square millimeters
Arm/Group | Ranibizumab Mono | PRP Mono | Ranibizumab+PRP
Number analyzed (Participants) | 33 | 32 | 33
square millimeters | -5.9 (12.7) | -0.7 (2.8) | -2.7 (3.9)
Statistical Analysis 1: Comparison: Ranibizumab Mono vs PRP Mono; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0081, ANCOVA; Least Squares Mean Difference = -2.4, 95% CI 2-sided [-4.2 to -0.6]
Statistical Analysis 2: Comparison: Ranibizumab Mono vs Ranibizumab+PRP; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.7494, ANCOVA; Least Squares Mean Difference = -0.3, 95% CI 2-sided [-2.0 to 1.5]
Statistical Analysis 3: Comparison: PRP Mono vs Ranibizumab+PRP; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0175, ANCOVA; Least Squares Mean Difference = 2.1, 95% CI 2-sided [0.4 to 3.9]

3. Secondary Outcome: Best Corrected Visual Acuity (BCVA) (ETDRS Letters) at EOCS
Description: BCVA was assessed using Early Treatment Diabetic Retinopathy Study (ETDRS)-like charts at a testing distance of 4 meters. A higher number of ETDRS letters may indicate better visual acuity. One eye (study eye) contributed to the analysis.
Time Frame: EOCS
Population: FAS; LOCF
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Ranibizumab Mono | PRP Mono | Ranibizumab+PRP
Number analyzed (Participants) | 35 | 35 | 36
letters | 84.4 (8.6) | 76.8 (17.0) | 78.9 (12.2)
Statistical Analysis 1: Comparison: Ranibizumab Mono vs PRP Mono; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0495, ANCOVA; Least Squares Mean Difference = 5.5, 95% CI 2-sided [0.0 to 11.0]
Statistical Analysis 2: Comparison: Ranibizumab Mono vs Ranibizumab+PRP; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.2767, ANCOVA; Least Squares Mean Difference = 3.0, 95% CI 2-sided [-2.5 to 8.5]
Statistical Analysis 3: Comparison: PRP Mono vs Ranibizumab+PRP; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.3641, ANCOVA; Least Squares Mean Difference = -2.5, 95% CI 2-sided [-7.9 to 2.9]

4. Secondary Outcome: Percentage of Patients With Change From Baseline in BCVA (ETDRS Letters) at EOCS
Description: BCVA was assessed using Early Treatment Diabetic Retinopathy Study (ETDRS)-like charts at a testing distance of 4 meters. No clinically relevant change was defined as <5 letters gain or loss. A higher positive change value may indicate a greater improvement in visual acuity. One eye (study eye) contributed to the analysis.
Time Frame: Baseline, EOCS
Population: FAS; LOCF
Measure: Number; unit: percentage of participants
Arm/Group | Ranibizumab Mono | PRP Mono | Ranibizumab+PRP
Number analyzed (Participants) | 35 | 35 | 36
percentage of participants
  ≥15 letters gain from Baseline at EOCS | 0.0 | 2.9 | 0.0
  ≥10 letters gain from Baseline at EOCS | 5.7 | 11.4 | 8.3
  ≥5 letters gain from Baseline at EOCS | 31.4 | 20.0 | 13.9
  No clinically relevant change from Baseline | 51.4 | 42.9 | 61.1
  ≥5 letters loss from Baseline at EOCS | 17.1 | 37.1 | 25.0
  ≥10 letters loss from Baseline at EOCS | 11.4 | 11.4 | 8.3
  ≥15 letters loss from Baseline at EOCS | 2.9 | 8.6 | 2.8
Statistical Analysis 1: Comparison: Ranibizumab Mono vs PRP Mono; ≥10 letters gain; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.4019, Regression, Logistic; Odds Ratio (OR) = 0.470, 95% CI 2-sided [0.080 to 2.749]
Statistical Analysis 2: Comparison: Ranibizumab Mono vs PRP Mono; ≥5 letters gain; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.2772, Regression, Logistic; Odds Ratio (OR) = 1.833, 95% CI 2-sided [0.614 to 5.471]
Statistical Analysis 3: Comparison: Ranibizumab Mono vs PRP Mono; No clinically relevant change; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.4731, Regression, Logistic; Odds Ratio (OR) = 1.412, 95% CI 2-sided [0.55 to 3.622]
Statistical Analysis 4: Comparison: Ranibizumab Mono vs PRP Mono; ≥5 letters loss; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.065, Regression, Logistic; Odds Ratio (OR) = 0.350, 95% CI 2-sided [0.155 to 1.068]
Statistical Analysis 5: Comparison: Ranibizumab Mono vs PRP Mono; ≥10 letters loss; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 1.000, Regression, Logistic; Odds Ratio (OR) = 1.000, 95% CI 2-sided [0.229 to 4.361]
Statistical Analysis 6: Comparison: Ranibizumab Mono vs PRP Mono; ≥15 letters loss; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.3261, Regression, Logistic; Odds Ratio (OR) = 0.314, 95% CI 2-sided [0.031 to 3.173]
Statistical Analysis 7: Comparison: Ranibizumab Mono vs Ranibizumab+PRP; ≥10 letters gain; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.6680, Regression, Logistic; Odds Ratio (OR) = 0.667, 95% CI 2-sided [0.104 to 4.253]
Statistical Analysis 8: Comparison: Ranibizumab Mono vs Ranibizumab+PRP; ≥5 letters gain; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0838, Regression, Logistic; Odds Ratio (OR) = 2.842, 95% CI 2-sided [0.870 to 9.283]
Statistical Analysis 9: Comparison: Ranibizumab Mono vs Ranibizumab+PRP; No clinically relevant change; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.4116, Regression, Logistic; Odds Ratio (OR) = 0.674, 95% CI 2-sided [0.263 to 1.729]
Statistical Analysis 10: Comparison: Ranibizumab Mono vs Ranibizumab+PRP; ≥5 letters loss; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.4197, Regression, Logistic; Odds Ratio (OR) = 0.621, 95% CI 2-sided [0.195 to 1.977]
Statistical Analysis 11: Comparison: Ranibizumab Mono vs Ranibizumab+PRP; ≥10 letters loss; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.6632, Regression, Logistic; Odds Ratio (OR) = 1.419, 95% CI 2-sided [0.294 to 6.856]
Statistical Analysis 12: Comparison: Ranibizumab Mono vs Ranibizumab+PRP; ≥15 letters loss; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.9839, Regression, Logistic; Odds Ratio (OR) = 1.029, 95% CI 2-sided [0.062 to 17.127]
Statistical Analysis 13: Comparison: PRP Mono vs Ranibizumab+PRP; ≥10 letters gain; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.6630, Regression, Logistic; Odds Ratio (OR) = 1.419, 95% CI 2-sided [0.294 to 6.858]
Statistical Analysis 14: Comparison: PRP Mono vs Ranibizumab+PRP; ≥5 letters gain; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.4941, Regression, Logistic — P-value was calculated as a point estimate; Odds Ratio (OR) = 1.550, 95% CI 2-sided [0.441 to 5.444]
Statistical Analysis 15: Comparison: PRP Mono vs Ranibizumab+PRP; No clinically relevant change; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.1259, Regression, Logistic; Odds Ratio (OR) = 0.477, 95% CI 2-sided [0.185 to 1.231]
Statistical Analysis 16: Comparison: PRP Mono vs Ranibizumab+PRP; ≥5 letters loss; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.2710, Regression, Logistic; Odds Ratio (OR) = 1.773, 95% CI 2-sided [0.640 to 4.913]
Statistical Analysis 17: Comparison: PRP Mono vs Ranibizumab+PRP; ≥10 letters loss; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.6632, Regression, Logistic; Odds Ratio (OR) = 1.419, 95% CI 2-sided [0.294 to 6.856]
Statistical Analysis 18: Comparison: PRP Mono vs Ranibizumab+PRP; ≥15 letters loss; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.3140, Regression, Logistic; Odds Ratio (OR) = 3.282, 95% CI 2-sided [0.325 to 33.171]

5. Secondary Outcome: Number of Patients With Change From Baseline in ETDRS Severity Grade of Diabetic Retinopathy (DR) at EOCS
Description: The severity level of diabetic retinopathy was determined using the ETDRS severity scale. However, in contrast to the original ETDRS severity scale, wide field fluorescein angiography images were used in addition to color fundus photography for identification of NVs and prior PRP treatment was not considered for determining the severity level. Eyes could be graded in the following classes: "DR absent" (10), "questionable DR" (14,15), "NPDR" (20-53), "mild PDR" (60-61), "moderate PDR" (65), "high risk PDR" (71-75), "advanced PDR" (81-85) and "cannot grade" (90). One eye (study eye) contributed to the analysis. No statistical analysis was conducted for ≥ 1 class deterioration or ≥ 2 class deterioration from Baseline at EOCS because ratios could not be calculated in case of zero frequencies in at least one of the three treatment groups.
Time Frame: Baseline, EOCS
Population: FAS. Only patients with both values at baseline and any post-baseline value were included.
Measure: Number; unit: participants
Arm/Group | Ranibizumab Mono | PRP Mono | Ranibizumab+PRP
Number analyzed (Participants) | 29 | 26 | 28
participants
  ≥ 1 class improvement from Baseline at EOCS | 10 | 9 | 13
  ≥ 2 class improvement from Baseline at EOCS | 2 | 2 | 5
  ≥ 1 class deterioration from Baseline at EOCS | 2 | 0 | 1
  ≥ 2 class deterioration from Baseline at EOCS | 0 | 0 | 0
Statistical Analysis 1: Comparison: Ranibizumab Mono vs PRP Mono; ≥ 1 class improvement from Baseline at EOCS; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.9918, Regression, Logistic; Odds Ratio (OR) = 0.994, 95% CI 2-sided [0.327 to 3.026]
Statistical Analysis 2: Comparison: Ranibizumab Mono vs Ranibizumab+PRP; ≥ 1 class improvement from Baseline at EOCS; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.3595, Regression, Logistic; Odds Ratio (OR) = 0.607, 95% CI 2-sided [0.209 to 1.765]
Statistical Analysis 3: Comparison: PRP Mono vs Ranibizumab+PRP; ≥ 1 class improvement from Baseline at EOCS; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.3787, Regression, Logistic; Odds Ratio (OR) = 0.611, 95% CI 2-sided [0.204 to 1.830]
Statistical Analysis 4: Comparison: Ranibizumab Mono vs PRP Mono; ≥ 2 class improvement from Baseline at EOCS; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.9097, Regression, Logistic; Odds Ratio (OR) = 0.889, 95% CI 2-sided [0.116 to 6.806]
Statistical Analysis 5: Comparison: Ranibizumab Mono vs Ranibizumab+PRP; ≥ 2 class improvement from Baseline at EOCS; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.2230, Regression, Logistic; Odds Ratio (OR) = 0.341, 95% CI 2-sided [0.060 to 1.925]
Statistical Analysis 6: Comparison: PRP Mono vs Ranibizumab+PRP; ≥ 2 class improvement from Baseline at EOCS; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.2792, Regression, Logistic; Odds Ratio (OR) = 0.383, 95% CI 2-sided [0.068 to 2.177]

6. Secondary Outcome: Change From Baseline in Central Subfield Thickness at EOCS
Description: Central subfield retinal thickness was assessed by a central reading center using Optical Coherence Tomography images. A positive change value may indicate disease progression. One eye (study eye) contributed to the analysis.
Time Frame: Baseline, EOCS
Population: FAS; LOCF. Only patients with both values at baseline and any post-baseline value were included.
Measure: Mean (Standard Deviation); unit: micrometer
Arm/Group | Ranibizumab Mono | PRP Mono | Ranibizumab+PRP
Number analyzed (Participants) | 32 | 31 | 31
micrometer | -6.0 (15.1) | 36.2 (55.9) | 17.6 (46.7)
Statistical Analysis 1: Comparison: Ranibizumab Mono vs PRP Mono; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0003, ANCOVA; Least Squares Mean Difference = -40.7, 95% CI 2-sided [-62.1 to -19.3]
Statistical Analysis 2: Comparison: Ranibizumab Mono vs Ranibizumab+PRP; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0357, ANCOVA; Least Squares Mean Difference = -22.9, 95% CI 2-sided [-44.2 to -1.6]
Statistical Analysis 3: Comparison: PRP Mono vs Ranibizumab+PRP; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.1034, ANCOVA; Least Squares Mean Difference = 17.8, 95% CI 2-sided [-3.7 to 39.3]

7. Secondary Outcome: Change From Baseline in Foveal Center Point Retinal Thickness at EOCS
Description: Foveal center point retinal thickness was assessed by a central reading center using Optical Coherence Tomography images. A positive change value may indicate disease progression. One eye (study eye) contributed to the analysis.
Time Frame: Baseline, EOCS
Population: FAS; LOCF. Only patients with both values at baseline and any post-baseline value were included.
Measure: Mean (Standard Deviation); unit: micrometer
Arm/Group | Ranibizumab Mono | PRP Mono | Ranibizumab+PRP
Number analyzed (Participants) | 32 | 31 | 31
micrometer | -4.7 (21.2) | 48.1 (83.7) | 25.5 (53.5)
Statistical Analysis 1: Comparison: Ranibizumab Mono vs PRP Mono; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0007, ANCOVA; Least Squares Mean Difference = -51.7, 95% CI 2-sided [-81.1 to -22.3]
Statistical Analysis 2: Comparison: Ranibizumab Mono vs Ranibizumab+PRP; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0542, ANCOVA; Least Squares Mean Difference = -28.9, 95% CI 2-sided [-58.4 to 0.5]
Statistical Analysis 3: Comparison: PRP Mono vs Ranibizumab+PRP; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.1288, ANCOVA; Least Squares Mean Difference = 22.8, 95% CI 2-sided [-6.7 to 52.3]

8. Secondary Outcome: Number of Ranibizumab Injections Until EOCS
Description: The total number of ranibizumab injections until EOCS was calculated. One eye (study eye) contributed to the analysis. No statistical analysis was conducted.
Time Frame: Baseline to EOCS
Population: Safety Set. This outcome measure was pre-specified for the ranibizumab mono and ranibizumab+PRP arms only.
Measure: Mean (Standard Deviation); unit: injections
Arm/Group | Ranibizumab Mono | PRP Mono | Ranibizumab+PRP
Number analyzed (Participants) | 35 | 35 | 36
injections | 5.2 (2.3) | NA (NA) — This outcome measure was pre-specified for the ranibizumab mono and ranibizumab+PRP arms only. | 5.0 (2.2)

9. Secondary Outcome: Number of PRP Laser Spots Until EOCS
Description: The total number of PRP laser spots from baseline until EOCS was calculated. One eye (study eye) contributed to the analysis. No statistical analysis was conducted.
Time Frame: Baseline to EOCS
Population: Safety Set. Only patients with at least 1 laser therapy until EOCS are included in the analysis. This outcome measure was pre-specified for the PRP and the ranibizumab+PRP arms only.
Measure: Mean (Standard Deviation); unit: PRP laser spots
Arm/Group | Ranibizumab Mono | PRP Mono | Ranibizumab+PRP
Number analyzed (Participants) | 35 | 35 | 36
PRP laser spots | NA (NA) — This outcome measure was pre-specified for the PRP and the ranibizumab+PRP arms only. | 1919.4 (673.1) | 1670.0 (568.4)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from time of informed consent until 4 weeks after the patient has stopped study participation (approximately 2 years).
Description: The Safety Set consisted of all randomized patients with at least one post-baseline safety assessment.
Groups:
- Ranibizumab Mono Until Month 12; PRP Mono Until Month 12; Ranibizumab+PRP Until Month 12: All visits up to Month 12 (which could lie after EOCS for patients who discontinued the core phase of the study)
- Ranibizumab Mono Month 12 to 24; PRP Mono Month 12 to 24; Ranibizumab+PRP Month 12 to 24: Non-interventional follow up phase
Arm/Group | Ranibizumab Mono Until Month 12 | PRP Mono Until Month 12 | Ranibizumab+PRP Until Month 12 | Ranibizumab Mono Month 12 to 24 | PRP Mono Month 12 to 24 | Ranibizumab+PRP Month 12 to 24
All-Cause Mortality (participants affected / at risk) | 1/35 | 1/35 | 2/36 | 0/28 | 0/20 | 0/25
Serious Adverse Events (participants affected / at risk) | 8/35 | 11/35 | 16/36 | 5/28 | 5/20 | 11/25
Other Adverse Events (participants affected / at risk) | 34/35 | 29/35 | 34/36 | 21/28 | 12/20 | 21/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab Mono Until Month 12 (N=35) | PRP Mono Until Month 12 (N=35) | Ranibizumab+PRP Until Month 12 (N=36) | Ranibizumab Mono Month 12 to 24 (N=28) | PRP Mono Month 12 to 24 (N=20) | Ranibizumab+PRP Month 12 to 24 (N=25)
ACUTE MYOCARDIAL INFARCTION (Non-ocular) (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
ATRIAL FIBRILLATION (Non-ocular) (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
CONGESTIVE CARDIOMYOPATHY (Non-ocular) (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
CORONARY ARTERY DISEASE (Non-ocular) (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
HEART VALVE STENOSIS (Non-ocular) (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
SUDDEN HEARING LOSS (Non-ocular) (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
ANTERIOR CHAMBER DISORDER (Right eye) (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
CATARACT (Left eye) (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
CATARACT (Right eye) (Eye disorders) | 0 | 1 | 0 | 1 | 0 | 0
DIABETIC RETINAL OEDEMA (Left eye) (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
DIABETIC RETINAL OEDEMA (Right eye) (Eye disorders) | 0 | 0 | 1 | 1 | 0 | 0
DIABETIC RETINOPATHY (Left eye) (Eye disorders) | 1 | 1 | 0 | 0 | 2 | 2
DIABETIC RETINOPATHY (Right eye) (Eye disorders) | 0 | 1 | 2 | 0 | 1 | 1
GLAUCOMA (Right eye) (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
MACULAR FIBROSIS (Left eye) (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
MACULAR FIBROSIS (Right eye) (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
MACULAR OEDEMA (Left eye) (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
OPEN ANGLE GLAUCOMA (Right eye) (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
RETINAL DETACHMENT (Left eye) (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
RETINAL HAEMORRHAGE (Both eyes) (Eye disorders) | 1 | 0 | 0 | 1 | 0 | 0
RETINAL HAEMORRHAGE (Right eye) (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
RETINAL NEOVASCULARISATION (Right eye) (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 1
VISUAL ACUITY REDUCED (Left eye) (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
VITREOUS ADHESIONS (Right eye) (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
VITREOUS HAEMORRHAGE (Left eye) (Eye disorders) | 1 | 1 | 1 | 0 | 0 | 1
VITREOUS HAEMORRHAGE (Right eye) (Eye disorders) | 1 | 2 | 0 | 0 | 0 | 2
ABDOMINAL PAIN (Non-ocular) (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
CHRONIC GASTRITIS (Non-ocular) (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
DENTAL CYST (Non-ocular) (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
DIARRHOEA (Non-ocular) (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
UMBILICAL HERNIA (Non-ocular) (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
CHEST PAIN (Non-ocular) (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
GENERAL PHYSICAL HEALTH DETERIORATION (Non-ocular) (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
NON-CARDIAC CHEST PAIN (Non-ocular) (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
PERIPHERAL SWELLING (Non-ocular) (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
GASTROENTERITIS (Non-ocular) (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
INFECTED SKIN ULCER (Non-ocular) (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
LOCALISED INFECTION (Non-ocular) (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
MENINGITIS (Non-ocular) (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
OSTEOMYELITIS (Non-ocular) (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
OSTEOMYELITIS CHRONIC (Non-ocular) (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
POSTOPERATIVE WOUND INFECTION (Non-ocular) (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
FRACTURED COCCYX (Non-ocular) (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
HUMERUS FRACTURE (Non-ocular) (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
HYPHAEMA (Right eye) (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
KIDNEY CONTUSION (Non-ocular) (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
MENISCUS INJURY (Non-ocular) (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
RIB FRACTURE (Non-ocular) (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
SPINAL FRACTURE (Non-ocular) (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
TENDON RUPTURE (Non-ocular) (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
BLOOD GLUCOSE FLUCTUATION (Non-ocular) (Investigations) | 0 | 0 | 1 | 0 | 1 | 0
DEHYDRATION (Non-ocular) (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
DIABETES MELLITUS (Non-ocular) (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 1
HYPERGLYCAEMIA (Non-ocular) (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0
HYPOGLYCAEMIA (Non-ocular) (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
OBESITY (Non-ocular) (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1
INTERVERTEBRAL DISC PROTRUSION (Non-ocular) (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
OSTEITIS (Non-ocular) (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
CHRONIC LYMPHOCYTIC LEUKAEMIA (Non-ocular) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
GASTRIC CANCER (Non-ocular) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
CEREBROVASCULAR ACCIDENT (Non-ocular) (Nervous system disorders) | 1 | 0 | 2 | 0 | 0 | 0
DIZZINESS (Non-ocular) (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
PREGNANCY (Non-ocular) (Pregnancy, puerperium and perinatal conditions) | 1 | 1 | 0 | 0 | 0 | 0
PSYCHIATRIC DECOMPENSATION (Non-ocular) (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
CHRONIC KIDNEY DISEASE (Non-ocular) (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
COUGH (Non-ocular) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
DYSPNOEA (Non-ocular) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
COLD SWEAT (Non-ocular) (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
DIABETIC FOOT (Non-ocular) (Skin and subcutaneous tissue disorders) | 0 | 1 | 3 | 0 | 0 | 0
DIABETIC MICROANGIOPATHY (Non-ocular) (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
HYPERTENSION (Non-ocular) (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Non-ocular) (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
PERIPHERAL ARTERY OCCLUSION (Non-ocular) (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
PERIPHERAL VENOUS DISEASE (Non-ocular) (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab Mono Until Month 12 (N=35) | PRP Mono Until Month 12 (N=35) | Ranibizumab+PRP Until Month 12 (N=36) | Ranibizumab Mono Month 12 to 24 (N=28) | PRP Mono Month 12 to 24 (N=20) | Ranibizumab+PRP Month 12 to 24 (N=25)
HYPOTHYROIDISM (Non-ocular) (Endocrine disorders) | 0 | 0 | 0 | 0 | 2 | 0
ABNORMAL SENSATION IN EYE (Right eye) (Eye disorders) | 0 | 2 | 0 | 0 | 0 | 0
BLEPHARITIS (Both eyes) (Eye disorders) | 1 | 0 | 2 | 0 | 0 | 0
CATARACT (Both eyes) (Eye disorders) | 3 | 1 | 1 | 0 | 0 | 1
CATARACT (Right eye) (Eye disorders) | 1 | 1 | 0 | 2 | 0 | 1
CONJUNCTIVAL HAEMORRHAGE (Left eye) (Eye disorders) | 3 | 0 | 3 | 1 | 0 | 0
CONJUNCTIVAL HAEMORRHAGE (Right eye) (Eye disorders) | 2 | 0 | 2 | 1 | 1 | 0
CONJUNCTIVITIS ALLERGIC (Both eyes) (Eye disorders) | 3 | 0 | 1 | 0 | 0 | 0
CORNEAL EROSION (Left eye) (Eye disorders) | 2 | 0 | 6 | 0 | 0 | 0
CORNEAL EROSION (Right eye) (Eye disorders) | 3 | 5 | 1 | 0 | 0 | 0
CYSTOID MACULAR OEDEMA (Right eye) (Eye disorders) | 0 | 2 | 2 | 0 | 0 | 0
DIABETIC RETINAL OEDEMA (Left eye) (Eye disorders) | 0 | 1 | 2 | 0 | 0 | 1
DIABETIC RETINAL OEDEMA (Right eye) (Eye disorders) | 0 | 0 | 6 | 0 | 0 | 0
DIABETIC RETINOPATHY (Both eyes) (Eye disorders) | 0 | 1 | 2 | 1 | 0 | 0
DIABETIC RETINOPATHY (Left eye) (Eye disorders) | 7 | 1 | 7 | 2 | 0 | 4
DIABETIC RETINOPATHY (Right eye) (Eye disorders) | 4 | 2 | 3 | 2 | 0 | 0
DRY EYE (Both eyes) (Eye disorders) | 3 | 2 | 2 | 1 | 0 | 1
EYE IRRITATION (Left eye) (Eye disorders) | 0 | 1 | 4 | 0 | 0 | 0
EYE IRRITATION (Right eye) (Eye disorders) | 0 | 0 | 3 | 0 | 0 | 0
EYE PAIN (Left eye) (Eye disorders) | 2 | 3 | 5 | 0 | 0 | 0
EYE PAIN (Right eye) (Eye disorders) | 3 | 1 | 6 | 1 | 0 | 0
FOREIGN BODY SENSATION IN EYES (Left eye) (Eye disorders) | 2 | 0 | 0 | 0 | 0 | 0
FOREIGN BODY SENSATION IN EYES (Right eye) (Eye disorders) | 2 | 0 | 2 | 0 | 0 | 0
GLARE (Right eye) (Eye disorders) | 0 | 2 | 0 | 1 | 0 | 0
IRIS NEOVASCULARISATION (Left eye) (Eye disorders) | 0 | 0 | 2 | 0 | 0 | 0
IRIS NEOVASCULARISATION (Right eye) (Eye disorders) | 0 | 1 | 3 | 0 | 0 | 1
LACRIMATION INCREASED (Left eye) (Eye disorders) | 0 | 0 | 3 | 0 | 1 | 0
LACRIMATION INCREASED (Right eye) (Eye disorders) | 1 | 1 | 2 | 0 | 0 | 0
MACULAR FIBROSIS (Left eye) (Eye disorders) | 3 | 1 | 0 | 1 | 0 | 0
MACULAR FIBROSIS (Right eye) (Eye disorders) | 1 | 2 | 3 | 0 | 0 | 0
MACULAR OEDEMA (Both eyes) (Eye disorders) | 0 | 2 | 2 | 2 | 0 | 1
MACULAR OEDEMA (Left eye) (Eye disorders) | 5 | 4 | 4 | 2 | 4 | 3
MACULAR OEDEMA (Right eye) (Eye disorders) | 3 | 8 | 4 | 5 | 1 | 4
OCULAR DISCOMFORT (Left eye) (Eye disorders) | 3 | 0 | 0 | 0 | 0 | 0
OCULAR HYPERAEMIA (Left eye) (Eye disorders) | 4 | 0 | 4 | 0 | 0 | 0
OCULAR HYPERAEMIA (Right eye) (Eye disorders) | 3 | 0 | 4 | 0 | 0 | 0
PUNCTATE KERATITIS (Both eyes) (Eye disorders) | 0 | 3 | 0 | 0 | 0 | 0
RETINAL CYST (Right eye) (Eye disorders) | 0 | 3 | 0 | 0 | 0 | 1
RETINAL EXUDATES (Left eye) (Eye disorders) | 2 | 2 | 0 | 0 | 0 | 0
RETINAL HAEMORRHAGE (Left eye) (Eye disorders) | 5 | 0 | 3 | 1 | 0 | 1
RETINAL HAEMORRHAGE (Right eye) (Eye disorders) | 3 | 1 | 3 | 1 | 0 | 2
RETINAL ISCHAEMIA (Left eye) (Eye disorders) | 1 | 0 | 2 | 1 | 0 | 1
RETINAL NEOVASCULARISATION (Both eyes) (Eye disorders) | 1 | 1 | 2 | 0 | 0 | 5
RETINAL NEOVASCULARISATION (Left eye) (Eye disorders) | 5 | 4 | 9 | 8 | 0 | 4
RETINAL NEOVASCULARISATION (Right eye) (Eye disorders) | 12 | 3 | 10 | 5 | 2 | 4
VISION BLURRED (Right eye) (Eye disorders) | 0 | 2 | 4 | 0 | 0 | 0
VISUAL ACUITY REDUCED (Both eyes) (Eye disorders) | 2 | 1 | 2 | 1 | 0 | 1
VISUAL ACUITY REDUCED (Left eye) (Eye disorders) | 5 | 3 | 12 | 2 | 1 | 1
VISUAL ACUITY REDUCED (Right eye) (Eye disorders) | 7 | 9 | 5 | 3 | 3 | 1
VISUAL IMPAIRMENT (Left eye) (Eye disorders) | 1 | 1 | 2 | 1 | 0 | 1
VITREOUS ADHESIONS (Right eye) (Eye disorders) | 2 | 2 | 0 | 1 | 0 | 0
VITREOUS DETACHMENT (Both eyes) (Eye disorders) | 0 | 2 | 0 | 0 | 0 | 0
VITREOUS FLOATERS (Left eye) (Eye disorders) | 3 | 1 | 0 | 0 | 0 | 1
VITREOUS FLOATERS (Right eye) (Eye disorders) | 0 | 0 | 2 | 0 | 0 | 0
VITREOUS HAEMORRHAGE (Left eye) (Eye disorders) | 6 | 6 | 5 | 4 | 2 | 4
VITREOUS HAEMORRHAGE (Right eye) (Eye disorders) | 4 | 7 | 5 | 3 | 1 | 7
DIARRHOEA (Non-ocular) (Gastrointestinal disorders) | 2 | 1 | 1 | 0 | 0 | 0
NAUSEA (Non-ocular) (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 0 | 1
TOOTHACHE (Non-ocular) (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0 | 0
VOMITING (Non-ocular) (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0 | 1
BRONCHITIS (Non-ocular) (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 2
GASTROENTERITIS (Non-ocular) (Infections and infestations) | 1 | 0 | 4 | 0 | 0 | 0
HORDEOLUM (Left eye) (Infections and infestations) | 2 | 2 | 0 | 1 | 0 | 0
INFLUENZA (Non-ocular) (Infections and infestations) | 0 | 2 | 2 | 0 | 0 | 0
NASOPHARYNGITIS (Non-ocular) (Infections and infestations) | 7 | 12 | 9 | 2 | 2 | 3
RHINITIS (Non-ocular) (Infections and infestations) | 2 | 1 | 1 | 0 | 0 | 0
SINUSITIS (Non-ocular) (Infections and infestations) | 0 | 2 | 2 | 0 | 0 | 2
CONTUSION (Non-ocular) (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 1 | 0 | 0
FALL (Non-ocular) (Injury, poisoning and procedural complications) | 1 | 3 | 0 | 0 | 0 | 0
FOOT FRACTURE (Non-ocular) (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0
PROCEDURAL PAIN (Both eyes) (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 0 | 0 | 0
PROCEDURAL PAIN (Left eye) (Injury, poisoning and procedural complications) | 0 | 2 | 4 | 0 | 0 | 0
RIB FRACTURE (Non-ocular) (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2
ROAD TRAFFIC ACCIDENT (Non-ocular) (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2
SCRATCH (Non-ocular) (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0
BLOOD CHOLESTEROL INCREASED (Non-ocular) (Investigations) | 0 | 0 | 1 | 3 | 1 | 0
BLOOD PRESSURE INCREASED (Non-ocular) (Investigations) | 0 | 1 | 0 | 2 | 0 | 0
BLOOD TRIGLYCERIDES INCREASED (Non-ocular) (Investigations) | 1 | 0 | 0 | 2 | 2 | 1
GLYCOSYLATED HAEMOGLOBIN INCREASED (Non-ocular) (Investigations) | 4 | 0 | 6 | 3 | 2 | 1
INTRAOCULAR PRESSURE INCREASED (Left eye) (Investigations) | 1 | 0 | 3 | 0 | 0 | 0
INTRAOCULAR PRESSURE INCREASED (Right eye) (Investigations) | 1 | 0 | 2 | 0 | 0 | 0
HYPERCHOLESTEROLAEMIA (Non-ocular) (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 1
ARTHRITIS (Non-ocular) (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0 | 0 | 0
PAIN IN EXTREMITY (Non-ocular) (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3 | 1 | 0 | 2
HEADACHE (Non-ocular) (Nervous system disorders) | 2 | 4 | 5 | 0 | 0 | 1
COUGH (Non-ocular) (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 3 | 0 | 0 | 0
DIABETIC FOOT (Non-ocular) (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0
HYPERTENSION (Non-ocular) (Vascular disorders) | 2 | 1 | 0 | 1 | 1 | 1
RETINAL ISCHAEMIA (Right eye) (Eye disorders) | 1 | 0 | 2 | 1 | 0 | 1
VITAMIN D DEFICIENCY (Non-ocular) (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0 | 0
BACK PAIN (Non-ocular) (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.